CLINICAL TRIAL: NCT05810987
Title: Remote Education Strategies Training Oncology Residents for End-of-Life Discussions (The RESTORED Study)
Brief Title: Remote Education Strategies Training Oncology Residents for End-of-Life Discussions
Acronym: RESTORED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14948
Record Dates: First submitted 2023-02-28; First posted 2023-04-13 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Oncology
Keywords: Communication, Serious Illness, Education, Palliative Care
MeSH Terms: conditions — Neoplasms; Communication | interventions — Restore polishing paste

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELMs and virtual SP encounters (Experimental): A virtual communication curriculum featuring electronic learning modules (ELMs) and skills sessions with standardized patients (SPs) along with coaching feedback.
  Interventions: Other: RESTORE; Behavioral: Medical Interaction and Coaching
- ELMs alone (Active Comparator): A virtual communication curriculum featuring electronic learning modules (ELMs) only.
  Interventions: Other: RESTORE

INTERVENTIONS:
Other: RESTORE — Virtual educational curriculum organized into the following modules:
  Module Specific Communication Strategies
  1. Introduction
  2. Preparing for and introducing a conversation [Consider personal bias /Building rapport /Ask permission]
  3. Assessing understanding [Avoid correcting /Open ended questions]
  4. Giving information [Give a warning shot /Using silence /Wish/worry/wonder]
  5. Explore goals [Reflective listening /Naming, validating emotion
  6. Summarizing and recommending a plan [Values-based recommendation /Aligning with goals /REMAP (Reframe, Expect emotion, Map goals, Align, Propose plan)]
Behavioral: Medical Interaction and Coaching — Skills sessions with standardized patients (SPs) along with coaching feedback.
  Arms: ELMs and virtual SP encounters

SUMMARY:
Difficult conversations are common in oncology practice and patient-centered communication is essential to care for individuals with cancer. Within oncology training programs, communication training is mostly unstructured observation and feedback in the clinic and many learners receive inadequate training. Currently, educational resources are limited, and residents have indicated a desire for more education on end-of-life communication skills. A formal communication curriculum could fill a gap and help to standardize teaching and evaluation.

The overall goal of this study is to establish an effective communication skills curriculum for oncology residents that can be delivered remotely and that addresses difficult conversations with cancer patients. Through this preliminary study, we will explore the feasibility of a randomized controlled trial comparing different training experiences to understand how best to help oncology residents develop strong end-of-life communication skills.

DETAILED DESCRIPTION:
Background:

Patient-centered communication is essential to care for individuals with cancer. High quality communication benefits patients, families, and clinicians. Proficiency in a variety of communication tasks is now a requirement within competency-based medical education (CBME) in Canada. Within oncology training programs, communication training is mostly unstructured observation and feedback in the clinic and many learners receive inadequate training. A formal communication curriculum could fill a gap and help to standardize teaching and evaluation, but current resources are limited.

Virtual care has been quickly adopted within oncology practice in the context of the COVID19 pandemic. This limits opportunities for direct observation of learners making assessment of communication skills more difficult. How best to teach communication skills in the context of virtual care is unclear. To mitigate current challenges, we will adapt two recognized educational tools, electronic learning modules (ELMs) and standardized patients (SPs), to create a novel virtual training strategy. Typically, SP skills sessions occur in person and effectiveness of SP encounters in a virtual care context has not been evaluated. Moreover, it is uncertain whether SPs are necessary for creation of psychological fidelity or improvement of transfer of communication skills. Thus, we aim to explore the relative impact of each component of a virtual communication curriculum. In this study, we will explore the feasibility of a randomized controlled trial comparing different training experiences.

Methods:

ELMs will be developed to teach communication skills for difficult conversations in oncology care. A framework for patient-centered communication and specific communication strategies will be introduced. Scenarios will be developed for virtual SP encounters related to each ELM. Virtual SP encounters will occur through the Zoom platform and include feedback from a remote faculty observer.

A randomized feasibility trial will be conducted. Consenting medical and radiation oncology residents in participating training programs (McMaster, University of Ottawa, University of Toronto) will be randomly assigned to complete the ELMs and virtual SP encounters (experimental arm) vs the ELMs alone (control arm). Video recorded simulated patient encounters will be conducted before and after the curricular activities. Recordings will be scored by trained assessors with multiple rating scales to evaluate communication skills of the learner. Standardized patients will also rate quality of physician communication with a patient-directed rating scale. This design will allow testing of our innovative educational interventions and exploration of the likelihood of success of a future RCT which will evaluate the impact of different training experiences. Outcome measures will include feasibility metrics such as recruitment, randomization, representativeness, adherence to intervention, and completeness of data collection. We will determine variance in scores on multiple rating scales within this study population to inform sample size of a future RCT. In addition, surveys completed pre- and post-intervention will assess change in self-efficacy rating and satisfaction with the learning experience.

Analysis:

The proposed sample size is 40 (20 per arm). This is based on achieving a 95% confidence interval (CI) of 60 to 85% around an estimated recruitment proportion of 75%. The primary outcome will be whether feasibility metrics meet criteria for success. Descriptive statistics with corresponding 95% CIs will summarize recruitment, adherence to study procedures, satisfaction and self-efficacy rating. For assessment of video recorded virtual simulated patient encounters, correlations between scores from different rating scales will be performed using Pearson's coefficient. Inter-rater reliability for rating scales will be done using Cohen's Kappa.

Conclusions:

If criteria for success are met among feasibility outcomes, a national RCT will follow to evaluate impact of virtual SPs added to the ELM curriculum. These novel educational resources simulate virtual care, a new paradigm that will likely persist beyond the pandemic. This is a scalable intervention which may standardize and strengthen communication training among oncology residency programs across Canada.

ELIGIBILITY:
Inclusion Criteria:

* Medical and radiation oncology residents and fellows at McMaster University, and medical oncology residents at the Universities of Ottawa and Toronto.
* Enrollment in a participating training program, ability to participate in study-related activities in English, access to internet and a video-enabled computer (either personal or institutional) to support study-related activities

Exclusion Criteria:

* Not enrolled in a participating training program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
COM-ON (Communication in Oncology) Checklist | 3 months
  Validated rating scale assessing general and specific communication skills in oncology. Items are rated on a five-point Likert scale ranging from 0 = ''Skill not demonstrated at all'' to 5 = ''Skill fully demonstrated'', with higher scores denoting higher quality communication.
QQPPI (Questionnaire on the Quality of Physician-Patient Interaction) | 3 months
  Validated patient-facing rating scale of for quality of physician communication. Items are rated on a five-point Likert scale ranging from 1 = ''I do not agree'' to 5 = ''I fully agree'', with higher scores denoting higher quality communication.
Assessment rubric for 'entrustable professional activities' (EPAs) | 3 months
  Medical interaction analysis rating scale as defined by the Royal College of Physicians and Surgeons of Canada. Items are rated on a five-point Likert scale ranging from 1 = ''I do not agree'' to 5 = ''I fully agree'', with higher scores denoting higher quality communication.
Global rating scale | 3 months
  Overall rating scale of quality of physician communication. Items are rated on a five-point Likert scale ranging from 1 = ''I do not agree'' to 5 = ''I fully agree'', with higher scores denoting higher quality communication.

SECONDARY OUTCOMES:
End-of-Life Professional Caregiver Survey (EPCS) | 3 months
  Validated instrument assessing educational needs relating to palliative care for interprofessional members of the healthcare team. Items are rated on a five-point Likert scale ranging from 1 (lowest level of skill) to 5 (greatest level of skill), with higher scores denoting a higher level of skill.
RESTORED Questionnaire | Immediately after the intervention
  Participant satisfaction with training intervention. Items are rated on a five-point Likert scale ranging from 1 = ''I do not agree'' to 5 = ''I fully agree'', with higher scores denoting higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Oren Levine, MD, Principal Investigator — McMaster University
Locations (1):
- Juravinski Cancer Centre - Hamilton Health Sciences, Hamilton, Ontario, Canada